CLINICAL TRIAL: NCT02453503
Title: Comparison of Triamcinolone Acetonide Mucoadhesive Film and Licorice Mucoadhesive Film Effect on the Duration and Symptoms of Lesions That Caused by Symptomatic Oral Lichen Planus
Brief Title: Comparison of Triamcinolone Acetonide Mucoadhesive Film and Licorice Mucoadhesive Film Effect on Lichen Planus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mehdi Nasr Isfahani, Director, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 394115
Record Dates: First submitted 2015-05-15; First posted 2015-05-25 (Estimated); Last update posted 2015-05-25 (Estimated); Status verified 2015-05

CONDITIONS: Oral Lichen Planus
Keywords: Lichen planus; Mucoadhesive film; licorice
MeSH Terms: conditions — Lichen Planus, Oral; Lichen Planus | interventions — Glycyrrhiza glabra extract; Triamcinolone Acetonide; Triamcinolone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Triamcinolone acetonide (Active Comparator): Triamcinolone acetonide mucoadhesive films 1 mg every 6 hours for two weeks.
  Interventions: Drug: Triamcinolone Acetonide
- Licorice (Experimental): Licorice mucoadhesive films 1 mg every 6 hours for two weeks.
  Interventions: Drug: Licorice

INTERVENTIONS:
Drug: Licorice — licorice mucoadhesive films evey 6 hours for two weeks
  Other Names: Aftogel
  Arms: Licorice
Drug: Triamcinolone Acetonide — Triamcinolone acetonide mucoadhesive films 1 mg every 6 hours for two weeks.
  Other Names: Triamcinolone
  Arms: Triamcinolone acetonide

SUMMARY:
Introduction :Oral lichen planus (OLP) is one of the most common disorders of the oral cavity which is basically a chronic and inflammated mucocutaneous .There is no cure for OLP currently. The main focus of treatment is to reduce the duration and severity of the symptoms. This study was designed to determine and compare the parameters of improvement in patient symptoms and lesions caused by oral lichen planus by using triamcinolone acetonide mucoadhesive film and licorice mucoadhesive film.

Methods and materials :The study was randomized by double-blind clinical trial . Patients with symptomatic OLP who referred to the Oral Medicine School of Dentistryin Medical Sciences in Isfahan University participated voluntarily. The patients were divided into two groups that were including 30 samples in each group. The first group was treated with triamcinolone mucoadhesive film and the second group were treated with licorice mucoadhesive film. Data were analyzed by using the Mann-Whitney test and t-test in SPSS software.

DETAILED DESCRIPTION:
Introduction OLP is a chronic and inflammatory disease that frequently involves the oral mucosa. Clinical symptoms of OLP are various from white keratotic lesions without pain to erosion and painful injury (1). OLP episodic symptoms range from pain and irritation of the mouth that can affect the normal function and causes physical and mental pressure to patients.OLP can be seen in two main forms of reticular and erosive. Erosive OLP have been seen as injured Arytmatozo that enclosed by keratotic striae .These lesions are often follow by episodic symptoms of pain and irritation to severe discomfort and can cause a major negative impact on performance of oral system and l quality of life .So, being aware of the Clinical symptoms and management of these lesions are very important for the clinician. (4,3,2,1)

Although, these lesions rarely are life-threatening , discomfort and pain associated with abnormal caloric intake lead to nervosa, dehydrated in short order and malnutrition. It also increases the risk of infection and reduce the quality of life in patients greatly.(2,3). The main treatment for symptomatic OLP is prescribing systemic or topical corticosteroids . (1,3) and its strong type like triamcinolone has been increasingly used in the treatment of OLP (4).

Lichen planus is a chronic mucocutaneous disease and relatively common in middle-aged that affected 2- 0.2% of the population. Men and women are almost equally affected. In the mouth, white bilatera lesions sometimes cause wound The most common clinical pattern is linear (9-5) .There is a limited study in the frequency and clinical forms of OLP.

It can be mention to Esmaeili etal study that patients in men and in fourth decades is most common and Hypertrophic and classic type are more and the type of reticular in oral lesions is more prevalent (10)and in another study by Khalili etal reported that the most common form of clinical lesion is ulcerated lesion and the average time spend 18.4 months, most commonly involving mucosa is the buccal and then the tongue and gums .White spots, lines Wickham and mucosal erythema are the most common clinical features of the lesion (11).

There is currently no cure for OLP. The main focus of treatment is to reduce the duration and severity of symptoms. The most common and acceptable treatment for symptomatic OLP lesions and systemic corticosteroids or topical is to modulate the host immune response .In mild to moderate lesions the main treatment is by topical corticosteroids such as clobetasol gel, betamethasone gel and triamcinolone ointment (2, 3, 12). Due to the persistence of the drug at the site of the lesion may be used new dosage form of mucoadhesive such as tablets or film. Films are from mucoadhesive drug delivery systems that have been used in the manufacture of mucoadhesive polymers and have received considerable attention in recent years .The films can be attached on the oral wound healing and cause to reduce pain and inflammatory diseases. (4, 13)

The Licorice plant have been used in traditional medicine for the treatment of aphthous ulcers, gastric ulcers, hepatitis C, cough, Asthma, Addison and skin diseases. Clinical pharmacology studies have shown that this herb also contains beneficial anti-inflammatory components, antiviral and antibacterial, antioxidant, anticancer and modifying the immune system is .Licorice contains a provision, glycyrrhetinic acid and glycyrrhizin which helps in healing wounds (14,15,16) In 2008, Martin et al. examined the effects of oral patch containing licorice extract (Licorice) for the treatment of aphthous ulcers and found positive effects on the size of the lesion and the patient's report of pain. (15) Chan et al., investigated palliative treatment of patients with symptomatic OLP such as steroids, Cyclosporine and topical retinoid in a systematic review and concluded that there are only weak evidence for the superiority of this treatment compared with placebo . The authors also expressed several studies has been faced with restrictions in which various compounds with potentially useful results on the OLP.

Conducted studies were not enough strong , the control group was small, making blind about the researcher or patient didn't do in them or have been made errors in designing the study. There would be special need to statistically powerful studies in order to determine the value of new compounds in the prevention or treatment of mucositis .(17)

The purpose of this study is to find a way to reduce pain and inflammation in patients with symptomatic OLP On the one hand and reduce the risk of infection, reduce the need for pain medication and ultimately improve the quality of life by using triamcinolone mucoadhesive films or licorice in this group of patients.

Methods and materials:

This study was a clinical trial and randomized as double-blind. Sampling was done randomly Patients with symptomatic OLP who referred to the Oral Medicine School of Dentistryin Medical Sciences in Isfahan University participated voluntarily.. In this study, patients with symptomatic OLP over 18 years both men and non-pregnant women enrolled in the study and . All patients were examined for dental Prophylaxis and oral hygiene and recommendations about compliance with oral health have been done for all patients . After filling written consent , the patients were divided into two groups randomly :first group I (n = 30) will be treated with triamcinolone Mucoadhesive film and the second group (n = 30) will be treated with licorice mucoadhesive film.

All patients underwent a complete dental examination and diagnosis of patients with oral lichen planus lesions initially marked by physical examination and conducted by interviewing with patients and then confirmed by histologic evaluation .The duration of treatment or recovery of lesions was two weeks as the weekly visits.

The Triamcinolone Mucoadhesive film with 1 mg was prepared and provided to patients in one group. And another group was given licorice mucoadhesive film by Afnogel brand name .The drug dose was determined three times a day after meals and before bed time that patients put it in the upper part of gum after eating and washing mouth and the patient can do common function like talking and eating and drinking within releasing the drug.

Severity and recovery rate of lesions were measured in each visit in accordance with the criteria that set in Buajeeb etal(18) from 0 to 5 degrees .The rate of pain in patients that created by Mucositis assessed by ruler and VAS method and it was given a number from 0 to 10 according to the rate of pain.

Injury or burning ,pain on waking, eating, drinking, talking, pain when swallowing, dry mouth, tingling or numbness after taking the studied medication and using the products containing caffeine, tobacco, and alcohol in the questionnaire registered by the patient .The compliance of patients were evaluated based on the returned mucoadhesive at the end of each week and based on the number of patients' visits to physicians. The patient withdrew from the study for any reason, pregnancy, drug interactions, compliance less than 70% patients about taking the medicine o has been done by referring to the doctor .All of the cases were collected and analyzed by the Mann-Whitney test.

ELIGIBILITY:
Inclusion Criteria:

* All patients over 18 years old
* All non pregnant women

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-01; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
VAS | 12 months
  Pain severity was measured by visual analogue scale : 0 for no pain and 10 for most painful experience